CLINICAL TRIAL: NCT02063646
Title: Effect of a Polyphenol-rich Food Supplement on Cognitive Function in Healthy Aging Adults: Randomized, Placebo-controlled, Double-blind Clinical Trial
Brief Title: Effect of a Polyphenol-rich Food Supplement on Cognitive Function in Healthy Aging Adults
Acronym: Neurophenol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurophenols Consortium (Other)
Collaborators: Activ'inside (Industry); Atrium Innovations (Industry); Fruit d'Or (Unknown); Laboratoire NutriNeuro Université de Bordeaux/INRA (Unknown); NutraCanada (Unknown); Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: INAF-2012-242
Record Dates: First submitted 2014-02-12; First posted 2014-02-14 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2014-10

CONDITIONS: Healthy Elderly
Keywords: polyphenols; memory; elderly

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): The placebo is a capsule with same appearance and organoleptic properties as the active product, containing no active component.
  Dose: 2 capsules per day, one capsule at least 1 hour after breakfast and one capsule at least one hour after dinner, with a glass of water.
  Interventions: Dietary Supplement: Placebo
- Polyphenol-rich extract (Experimental): The test product is a food supplement named Neurophenol. It is presented as a hard-shell capsule containing polyphenol-rich extracts.
  Dose: 2 capsules per day, one capsule at least 1 hour after breakfast and one capsule at least one hour after dinner, with a glass of water.
  Interventions: Dietary Supplement: Polyphenol-rich extract

INTERVENTIONS:
Dietary Supplement: Polyphenol-rich extract — Two groups, each of 102 volunteers, are studied. For 24 weeks, one group of volunteers will consume the active product (polyphenol-rich extract) while the other one will consume the placebo product.
  Arms: Polyphenol-rich extract
Dietary Supplement: Placebo — The placebo is a capsule with same appearance and organoleptic properties as the active product, containing no active component.
  Two groups, each of 102 volunteers, are studied. For 24 weeks, one group of volunteers will consume the active product (polyphenol-rich extract) while the other one will consume the placebo product.
  Arms: Placebo

SUMMARY:
Several preliminary studies have shown that diet can have beneficial effects on cognitive decline. Among food shown to have such effects are some polyphenols from selected botanicals.

Preclinical studies have concluded that polyphenols play a role in moderation of oxidative stress and inflammation, increased neuronal signaling, and improved metabolic function among other effects. Noteworthy, a positive and statistically significant association between the midlife level of polyphenol intake and cognitive function assessed 13 years later was found in a cohort of 2574 adults.

Several mechanisms may be involved in these positive effects of food polyphenols on cognitive function in older adults: experimental studies suggest that polyphenols display neuroprotective effects, enhancement of the neuronal function, stimulation of brain flow and inducing neurogenesis, and might prevent age-related damage to the central nervous system through their antioxidant and anti-inflammatory activities.

Based on these promising results, a food supplement from botanicals offering complementary polyphenol profile was developed. This food supplement is aimed to aid at maintenance of cognitive function in older adults.

DETAILED DESCRIPTION:
This project aims to investigate the effects of 6 months supplementation with a polyphenol-rich supplement vs. placebo to consume daily on human cognitive function. Polyphenol-rich supplement and placebo will be provided as capsules matched for appearance.

The study will be conducted as a randomized, double-blind, parallel-groups (2 arms) placebo-controlled, multicentre interventional design. Two groups, each of 102 volunteers, are studied. One group of volunteers will consume the polyphenol-rich product while the other one will consume the placebo product.

Each volunteer will be seen for 3 visits at the investigational site, will have 2 follow-up calls and mid-term dietary survey. Baseline and follow-up visit will include cognitive assessment with the CANTAB battery. CANTAB tests will cover several aspects of memory: visio-spatial learning and episodic memory, verbal recognition memory and visio-spatial working memory. Moreover, psychological and mood components will be evaluated (mnesic complaint, depression, fatigue). Physical activity and food habits will also be recorded. Finally, biological parameters will be assessed (lipid profile, glycemia, insulinemia, CRPus, thyroid stimulating hormone, transthyretin, plasma level of phenolic compounds).

ELIGIBILITY:
Inclusion Criteria:

* Independent subjects, living at home;
* Body Mass Index (BMI) 20-30 kg/m2 (limits included);
* 26 < MMSE score ≤ 29
* Logical memory subtest of the Wechsler Memory Scale (16-69 years battery) sub-scores complying with the following:

  * Immediate recall score < 29;
  * Delayed recall score < 16;

Exclusion Criteria:

* Evidence of actual major depressive disorder according to the module A of the Mini International Neuropsychiatric Interview (MINI);
* Subject consuming food supplements likely to have an effect on memory;
* High physical activity practice;
* Restrictive or unbalanced diet (hypocaloric, vegetarian, vegan, …) self-declared at V0;
* Diabetes;
* Cardiovascular disease diagnosed within less than 2 years, with the following exceptions: subjects with controlled (medicated) high blood pressure and/ or controlled (medicated) can be included;
* Personal history of Cerebrovascular Accident (CVA);
* Unbalanced thyroid disease;
* Anti-depressant treatment stopped since less than 3 months or still ongoing;
* Personal history of schizophrenia or other psychiatric disorders;
* Ongoing neuroleptic treatment;
* Uncorrected visual or auditory dysfunction (according to the volunteer's self-declaration);
* History of moderate to severe traumatic brain injury and / or intracranial surgery;
* Life threatening pathology (such as cancer) in remission for less than 1 year or still ongoing;
* General anesthesia in the last 6 months or planned in the next 6 months;
* Documented food allergy(ies), namely to one of the components of the study product;
* Psychological or linguistic incapability to sign the informed consent.

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
CANTAB - Paired Associate Learning test (PAL) | 24 weeks

SECONDARY OUTCOMES:
CANTAB - Verbal Recognition Memory (VRM) | 24 weeks
CANTAB - Spatial Span test (SSP) | 24 weeks
CANTAB - Reverse Spatial Span test (Reverse SSP) | 24 weeks
Wechsler Memory Scale - Logical memory subtest | 24 weeks
McNair scale | 24 weeks
Geriatric Depression Scale | 24 weeks
Mini-Mental State Examination | 24 weeks
Multidimensional Fatigue Inventory (MFI-20) | 24 weeks

OTHER OUTCOMES:
Lipid profile | 24 weeks
Insulinemia and glycemia | 24 weeks
Inflammatory markers | 24 weeks
Hormones | 24 weeks
Urinary polyphenols | 24 weeks
Fatty acid profile in erythrocyte membranes | 24 weeks
Retinol Binding Protein and Transtyretin | 24 weeks
Nuclear receptor expression in mononuclear cells | 24 weeks
Gene expression in mononuclear cells by microarray approach | 24 weeks
Epigenetic markers | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carol Hudon, Ph.D., Principal Investigator — Laval University; Véronique Pallet, Ph.D., Principal Investigator — Laboratoire NutriNeuro Université de Bordeaux/INRA; Catherine Bégin, Ph.D., Principal Investigator — Laval University
Locations (2):
- INAF (Institute of nutrition and functionnal foods), Québec, Quebec, Canada
- Biofortis, Saint-Herblain, France

REFERENCES:
- [Background] Krikorian R, Boespflug EL, Fleck DE, Stein AL, Wightman JD, Shidler MD, Sadat-Hossieny S. Concord grape juice supplementation and neurocognitive function in human aging. J Agric Food Chem. 2012 Jun 13;60(23):5736-42. doi: 10.1021/jf300277g. Epub 2012 Apr 9. PMID 22468945
- [Background] Kesse-Guyot E, Fezeu L, Andreeva VA, Touvier M, Scalbert A, Hercberg S, Galan P. Total and specific polyphenol intakes in midlife are associated with cognitive function measured 13 years later. J Nutr. 2012 Jan;142(1):76-83. doi: 10.3945/jn.111.144428. Epub 2011 Nov 16. PMID 22090468
- [Background] Rossi L, Mazzitelli S, Arciello M, Capo CR, Rotilio G. Benefits from dietary polyphenols for brain aging and Alzheimer's disease. Neurochem Res. 2008 Dec;33(12):2390-400. doi: 10.1007/s11064-008-9696-7. Epub 2008 Apr 16. PMID 18415677
- [Background] Spencer JP, Vauzour D, Rendeiro C. Flavonoids and cognition: the molecular mechanisms underlying their behavioural effects. Arch Biochem Biophys. 2009 Dec;492(1-2):1-9. doi: 10.1016/j.abb.2009.10.003. Epub 2009 Oct 12. PMID 19822127
- [Background] Vauzour D, Vafeiadou K, Rodriguez-Mateos A, Rendeiro C, Spencer JP. The neuroprotective potential of flavonoids: a multiplicity of effects. Genes Nutr. 2008 Dec;3(3-4):115-26. doi: 10.1007/s12263-008-0091-4. PMID 18937002
- See also: Click this link for more information about this study — http://www.neurophenols.org
- See also: Laboratoire NutriNeuro INRA-Université de Bordeaux — http://www6.bordeaux-aquitaine.inra.fr/nutrineuro